CLINICAL TRIAL: NCT05518045
Title: An Open-Label, Dose-Escalation and Dose-Expansion Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Efficacy of LM-108 for Injection as Monotherapy or in Combination With Antitumor Therapies in Patients With Advanced Solid Tumors
Brief Title: A Study of LM-108 as Monotherapy or in Combination With Antitumor Therapies in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM108-01-103
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LM-108 Dose Escalation (Experimental)
  Interventions: Drug: LM-108
- LM-108 Dose Expansion (Experimental)
  Interventions: Drug: LM-108
- LM-108 combination dose expansion (Experimental)
  Interventions: Drug: LM-108; Drug: Toripalimab

INTERVENTIONS:
Drug: LM-108 — Administered intravenously
Drug: Toripalimab — Administered intravenously
  Arms: LM-108 combination dose expansion

SUMMARY:
A Phase I/II, Open-Label, Dose-Escalation and Dose-Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Efficacy of LM-108, an Anti-CCR8 Monoclonal Antibody, as Monotherapy or in Combination with Antitumor Therapies in Patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
2. Histological or cytological confirmation of recurrent or refractory advanced solid tumours, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
3. At least one measurable disease for expansion cohorts per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
4. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose.

Exclusion Criteria:

1. Have received anti-CCR8 drug treatment or other clinical study drug or treatment not on the market within 28 days prior to the first dose.
2. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
3. Subjects with uncontrolled tumor-related pain.
4. Subjects with known brain metastases.
5. Uncontrollable clinical third luminal effusion.
6. Known history of autoimmune disease.
7. Use of any live attenuated vaccines within 28 days.
8. Have severe cardiovascular disease.
9. Uncontrolled or severe illness.
10. History of immunodeficiency disease.
11. Active malignancies which are likely to require the treatment.
12. Child-bearing potential female.
13. Have psychiatric illness or disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase I Dose Escalation:Incidence of adverse events (AEs) | 152 Weeks
Phase I Dose Escalation:Incidence of dose-limiting toxicity (DLT) | 152 Weeks
Phase I Dose Escalation:Incidence of serious adverse event (SAE) | 152 Weeks
Phase I Dose Escalation:Incidence of clinical significant in laboratory examinations, including hematology, urinalysis, blood biochemistry, coagulation tests and thyroid function. | 152 Weeks
Phase II Dose Expansion Cohort:Objective Response Rate (ORR) Evaluated by Researchers Based on RECIST v1.1 | 152 Weeks

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) for LM-108 | 152 Weeks
PK Parameter: Time of Maximum Observed Concentration (Tmax) for LM-108 | 152 Weeks
PK Parameter: Area Under the Concentration-time Curve (AUC) for LM-108 | 152 Weeks
PK Parameter: Steady State Maximum Concentration (Cmax,ss) | 152 Weeks
PK Parameter: Steady State Minimum Concentration (Cmin, ss) | 152 Weeks
PK Parameter: Systemic Clearance at Steady State (CLss) | 152 Weeks
PK Parameter: Accumulation Ratio (Rac) | 152 Weeks
PK Parameter: Elimination Half-life (t 1/2) | 152 Weeks
PK Parameter: Volume of Distribution at Steady-State (Vss) | 152 Weeks
PK Parameter: Degree of Fluctuation (DF) | 152 Weeks
Incidence of anti-drug antibodies to LM-108 | 152 Weeks
Phase I Dose Escalation：Preliminary anti-tumor activity：Objective Response Rate,Duration of Response, Disease Control Rate,Progression-Free Survival,and Overall Survival evaluated according to the Response Evaluation Criteria in Solid Tumors (RECISTv1.1) | 152 Weeks
Phase I Dose Escalation：Correlation between biomarker expression levels (FoxP3, PD-L1, CCR8, CD8) and the anti-tumor activity of LM-108 as monotherapy or in combination with toripalimab. | 152 Weeks
Phase II Dose Expansion Cohort:Antitumor Activity: Duration of Response (DOR), Disease Control Rate (DCR), Progression-Free Survival (PFS), and Overall Survival (OS) evaluated by investigators based on RECIST v1.1; | 152 Weeks
Phase II Dose Expansion Cohort:Objective Response Rate (ORR), DOR, DCR, and PFS evaluated by the Independent Review Committee (IRC) based on RECIST v1.1 | 152 Weeks
Phase II Dose Expansion Cohort:Incidence of adverse events (AEs) | 152 Weeks
Phase II Dose Expansion Cohort:Incidence of serious adverse event (SAE) | 152 Weeks
Phase II Dose Expansion Cohort:Incidence of clinical significant in laboratory examinations, including hematology, urinalysis, blood biochemistry, coagulation tests and thyroid function. | 152 Weeks
Phase II Dose Expansion Cohort:Correlation between biomarker expression levels (FoxP3, PD-L1, CCR8, CD8) and the anti-tumor activity of LM-108 as monotherapy or in combination with anti-tumor therapies. | 152 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No